CLINICAL TRIAL: NCT05612295
Title: Effect of Mindfulness-Based Intervention on Endurance Performance Under Pressure and Performance-Relevant Mental Attributes an Interdisciplinary Perspective
Brief Title: Mindfulness-Based Peak Performance, Endurance Performance Under Pressure, Performance-relevant Mental Attributes
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan Normal University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PACNL_MBPP_Stress
Record Dates: First submitted 2022-11-01; First posted 2022-11-10 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-11

CONDITIONS: Mindfulness; Sport Performance; Neurocognitive Function; Stress
Keywords: mindfulness intervention; sport performance under pressure; Neurocognitive function

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- MBPP group (Experimental): The Mindfulness-based Peak Performance (MBPP) program consists of eight 60-min training sessions, once weekly for 8 weeks, which aim to enhance human performance.
  Interventions: Behavioral: MBPP
- Self-talk group (Active Comparator): The self-talk intervention serving as the active control group will be included in the current trial. In line with the MBPP intervention, the self-talk intervention is also designed to enhance athletic performance, and will consist of eight 60-min meaningful sessions, once per week for eight weeks.
  Interventions: Behavioral: Self-talk
- Waiting-list control (No Intervention): The participants in waiting-list control group are advised to maintain their everyday lifestyles and regular training. Once the participants in WC finish the experiment, they will be invited to participate in one of the 8-week interventions (i.e., MBPP or ST) based upon their preference.

INTERVENTIONS:
Behavioral: MBPP — MBPP program consist of three fundamental principles (i.e., attention monitoring, acceptance, sport-specific rationale) and six performance-related core mental attributes including three behavioral and three neurocognitive components.
  Each session will start with a brief homework discussion and recap of the preceding session, and instructors will deliver a topic-related brief story or group activity to participants, followed by a theoretical introduction and practice of mindfulness. Finally, at the end of each session, instructors will guide participant to discuss mindfulness applications related to specific sports performances. At the end of the session, participants will be assigned homework to increase the effectiveness of MBPP, and participants will be encouraged to practice daily for at least 10-15 min between the sessions.
  Other Names: Mindfulness-based intervention
  Arms: MBPP group
Behavioral: Self-talk — self-talk sessions include: Session 1 & 2. The concepts, types, and the importance of self-talk will be introduced; Session 3. Researchers, coaches and the athletes will work together to design syntactically recognizable, concise, and clear sport-specific instructional scripts for specific sports performance (e.g., running); Session 4. practice of sport-specific instructional self-talk; Session 5. researchers, coaches and the athletes will work together to design syntactically recognizable, concise, and clear sport-specific motivational self-talk scripts for specific sports performances; Session 6. practice of sport-specific motivational self-talk; and Session 7 & 8. general practice for learned self-talk techniques.
  Arms: Self-talk group

SUMMARY:
The primary aim of this study is to conduct a well-designed trial to investigate the effect of an MBI program entitled Mindfulness-based Peak Performance (MBPP) on endurance performance under pressure from an interdisciplinary approach of sport psychology, sports training, and cognitive neuroscience. The secondary aim is to examine the effect of MBPP program on performance-relevant mental attributes in behavioral and neurocognitive assessments.

The present study hypothesizes that the MBPP and self-talk groups will improve performance under pressure, but MBPP is expected to show greater improvement than ST. Additionally, we expect the MBPP will improve the relevant mental attributes.

DETAILED DESCRIPTION:
Considering that increased competition levels are typically accompanied by elevated stress and anxiety, athletes' ability to cope with stress has gained even more importance in recent years. Growing evidence has demonstrated the effectiveness of mindfulness in reducing stress and enhancing athletic performance; however, its effectiveness remains a matter of debate and limitations due to absence of more rigorous designs, ecological validity, and randomized controlled trials.

Accordingly, the current trial, entitled Mindfulness-based Peak Performance (MBPP), will take an interdisciplinary approach (e.g., sport psychology, sports training, and cognitive neuroscience), to more definitively examine whether a tailored mindfulness-based intervention (MBI) affects athletic performance under pressure and relevant mental attributes.

Specifically, this study is an 8-week, three-arm, randomized controlled trial (RCT), and eligible participants will be randomly assigned into (1) an MBPP group (MBPP), (2) a self-talk group (ST), and (3) a wait-list control group (WC). The primary outcomes (e.g., endurance performance under pressure, performance-relevant mental attributes) and secondary outcomes (e.g., dispositional mindfulness, sports psychological skills) will be assessed before and after intervention.

The MBPP and ST are expected that will improve performance under pressure, but MBPP might show greater improvement than ST. Additionally, MBPP is expected that will improve performance-relevant mental attributes. The results from this trial might provide rigorous evidence and insight into MBI application in the sports context.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 30 years
* Normal or corrected-to-normal 20/20 vision
* No red-green color blindness
* Able to speak and read Chinese
* Physical Activity Readiness Questionnaire (PAR-Q) score = 0
* With one of the designated sport proficiencies (i.e., middle-long running, marathon, triathlon)
* No previous major experience in mindfulness-related training (e.g., meditation or Tai Chi)
* Provide informed consent

Exclusion Criteria:

* Diagnosed or self-reported cognitive problems
* The diagnosed or self-reported physical disease (e.g., untreated hypertension and chronic heart disease, stroke, brain tumor, musculoskeletal disorders, other exercise contradictions)
* Diagnosed or self-reported major psychiatric illness (e.g., major depression, schizophrenia)
* History of alcohol or drug abuse
* Unwillingness to be randomized to one of the three groups
* Currently participating in another study trial

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2023-12-31 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Endurance performance: Change in time to exhaustion | 30 minutes each at the Baseline-Assessment and at the Post-Assessment
  Time to exhaustion (TTE) will be one of the measured variables of endurance performance and be evaluated via a graded exercise test (GXT) on a motor-driven treadmill.
Endurance performance: Change in maximum oxygen consumption | 30 minutes each at the Baseline-Assessment and at the Post-Assessment
  Maximum oxygen consumption (VO2max) will be one of the measured variables of endurance performance and be evaluated via a computerized indirect calorimetry system throughout the whole graded exercise test (GXT) on a motor-driven treadmill.
Endocrine stress responses | 1 minutes for each sampling
  Before and after pressure manipulation, and after endurance performance measure, stress responses of endocrine assessments will be assessed. Specifically, salivary cortisol (sCort) and salivary alpha-amylases (sAA) will be collected using the commercially available sampling devices.
Subjective stress responses | 5 minutes for each assessment
  The participants' subjective perception of stress will be assessed via the Chinese version of the State-Trait Anxiety Inventory (C-STAI) (Wang and Chung, 2016) modified from the original version of STAI (Spielberger et al., 1971). The state subscale of the STAI will be the index of state anxiety influenced by pressure manipulation.
Change in emotion regulation | 10 minutes each at the Baseline-Assessment and at the Post-Assessment
  The Chinese version of the Difficulties in Emotion Regulation Scale (C-DERS) modified from DERS (Gratz and Roemer, 2004) will be used to assess emotional regulation. C-DERS is a 36-item self-reported questionnaire to measure the six facets of emotional regulation (i.e., awareness, clarity, impulse, goal, non-acceptance, and strategies). Items are rated on a 5-point Likert scale from 1 (almost never) to 5 (almost always).
Engagement | 5 minutes at the Post-Assessment
  Participants' engagement will be an adherence score calculated by addition of the Z scores for overall participant attendance of MBPP/ST sessions and a Z score for overall participant minutes spent on home practice, then divided by the total Z scores. Researchers will record the attendance of each participant in MBPP or ST programs.
Executive function: Change in reaction time | 30 minutes each at the Baseline-Assessment and at the Post-Assessment
  The executive function in terms of reaction time will be assessed by the computerized Stroop Test. The types of trials are the three Chinese color words printed in one of the three types of color. Based on the combination of words and the pixels of the color, there are three types of trials: (1) congruent trials: the stimuli in which the color of the word corresponds to the semantic meaning of the word; (2) incongruent trials: the stimuli in which the paint color of the word is inconsistent with the semantic meaning of the word; and (3) neutral trials: the colored squared.
Executive function: Change in accuracy | 30 minutes each at the Baseline-Assessment and at the Post-Assessment
  The executive function in terms of accuracy will also be assessed by the computerized Stroop Test. The types of trials are the three Chinese color words printed in one of the three types of color. Based on the combination of words and the pixels of the color, there are three types of trials: (1) congruent trials: the stimuli in which the color of the word corresponds to the semantic meaning of the word; (2) incongruent trials: the stimuli in which the paint color of the word is inconsistent with the semantic meaning of the word; and (3) neutral trials: the colored squared.
Change in attention | 30 minutes each at the Baseline-Assessment and at the Post-Assessment
  The attention will be measured by event-related potential while Stroop Test.
Change in brain resting state | 8 minutes each at the Baseline-Assessment and at the Post-Assessment
  The frequency domain of electroencephalography (EEG) will also be recorded during the resting state at baseline and post-intervention.

SECONDARY OUTCOMES:
General dispositional mindfulness | 5 minutes each at the Baseline-Assessment and at the Post-Assessment
  The general dispositional mindfulness will be assessed by Chinese version of the Mindful Attention Awareness Scale (C-MAAS)(Chang et al., 2011), which is modified from the original Mindful Attention Awareness Scale (MAAS; Brown & Ryan, 2003). Higher scores reflect higher levels of general dispositional mindfulness.
Athletic dispositional mindfulness | 5 minutes each at the Baseline-Assessment and at the Post-Assessment
  Athletic mindfulness will be measured by the Athlete Mindfulness Questionnaire (AMQ; Zhang et al., 2017). Higher scores reflect higher levels of athletic dispositional mindfulness.
Athletic psychological skills | 5 minutes each at the Baseline-Assessment and at the Post-Assessment
  Athletic psychological skill levels will be assessed using the Athletic Psychological Skill Inventory (APSI) (Chiou and Chi, 2001), which is a modified Chinese version of Athletic Coping Skills Inventory-28 (ACSI-28; Smith et al., 1995).

CONTACTS AND LOCATIONS:
Overall Officials: Yu-Kai Chang, Ph.D., Study Director — Department of Physical Education and Sport Sciences, National Taiwan Normal University
Locations (1):
- Department of Physical Education and Sport Sciences, National Taiwan Normal University, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No
Data are available upon request.

REFERENCES:
- [Derived] Chang YK, Gill DL, Creswell JD, Chen DT, Lin CY, Chu CH, Nien JT. Effect of mindfulness-based intervention on endurance performance under pressure and performance-relevant mental attributes, an interdisciplinary perspective: Protocol for a Mindfulness-Based Peak Performance (MBPP) trial. Contemp Clin Trials. 2023 Jun;129:107175. doi: 10.1016/j.cct.2023.107175. Epub 2023 Apr 5. PMID 37028503